CLINICAL TRIAL: NCT01245842
Title: Osteoarthritis Care in Primary Health: Hand Exercises and Telephone Counselling for Hand OA - a Randomized Controlled Trial
Brief Title: The Hand Osteoarthritis Exercise Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Principal Investigator, Nina Osteras, Principal Investigator, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 100286_1
Record Dates: First submitted 2010-11-19; First posted 2010-11-23 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Hand Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Usual care (No Intervention)
- Exercise group (Experimental)
  Interventions: Other: Hand exercise program

INTERVENTIONS:
Other: Hand exercise program — Hand exercise program three times/week for 12 weeks. In total four group sessions, otherwise home based. Weekly telephone calls from experienced physiotherapist/occupational therapist addressing adjustments of the exercise program and encouragement of program adherence.
  Arms: Exercise group

SUMMARY:
The purpose of this study is to evaluate the effect of a hand exercise intervention on function and osteoarthritis symptoms in persons with hand osteoarthritis .

DETAILED DESCRIPTION:
Hand osteoarthritis (OA) is one of the most prevalent musculoskeletal diseases in an adult population. The disease may have large influences on an individual's function, health related quality of life and participation in the society. In recently published clinical guidelines for management, non-pharmacological approaches are considered as core treatments.

Several studies have demonstrated that exercise may reduce pain and improve function in persons with knee OA, and a similar effect is suggested for hip OA. Regarding effect of exercises in hand OA, available research results are limited, and randomised controlled trials (RCT) of good quality are needed.

ELIGIBILITY:
Inclusion Criteria:

* The American College of Rheumatology (ACR) classification criteria for clinical hand osteoarthritis
* FIHOA ≥ 5 at pre-baseline
* The persons must have a telephone

Exclusion Criteria:

* Persons with cognitive dysfunction
* Persons who do not understand Norwegian language
* Persons with inflammatory rheumatic diseases (e.g. rheumatoid arthritis, ankylosing spondylitis) or cancer
* Persons that have recently experienced severe trauma
* Persons that have recently gone through OA surgery or other major surgery

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The functional index for hand osteoarthritis (FIHOA) | 6 months
Patient specific function scale (PSFS) | 6 months

SECONDARY OUTCOMES:
Hand joint pain (Numeric rating scale, 0-10) | 6 months
Hand joint stiffness (Numeric rating scale, 0-10) | 6 months
Fatigue (numeric rating scale, 0-10) | 6 months
Patient global assessment of disease activity (Numeric rating scale, 0-10) | 6 months
Exercise self-efficacy | 6 months
Health related quality of life (15D) | 6 months
Self-reported work ability and sick leave | 6 months
Self-reported health care utilisation | 6 months
Grip strength (JAMAR) | 6 months
Grip size | 6 months
Hand functioning (The Moberg Pick Up Test) | 6 months
Global assessment of change of hand problem | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nina Østerås, PT, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (1):
- Physiotherapy and Occupational Therapy Service Centre, Ullensaker Municipality, Jessheim, Norway

REFERENCES:
- [Derived] Osteras N, Hagen KB, Grotle M, Sand-Svartrud AL, Mowinckel P, Kjeken I. Limited effects of exercises in people with hand osteoarthritis: results from a randomized controlled trial. Osteoarthritis Cartilage. 2014 Sep;22(9):1224-33. doi: 10.1016/j.joca.2014.06.036. Epub 2014 Jul 5. PMID 25008206
- [Derived] Osteras N, Hagen KB, Grotle M, Sand-Svartrud AL, Mowinckel P, Aas E, Kjeken I. Exercise programme with telephone follow-up for people with hand osteoarthritis - protocol for a randomised controlled trial. BMC Musculoskelet Disord. 2014 Mar 14;15:82. doi: 10.1186/1471-2474-15-82. PMID 24629063